CLINICAL TRIAL: NCT01254864
Title: Maximal Androgen Depletion Followed by Randomization of Maximal Androgen Ablation With Molecular Targeted Therapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Janssen Scientific Affairs, LLC (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0070; NCI-2011-00267 (Registry Identifier: NCI CTRP-Clinical Trials Registry)
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Castrate resistant prostate cancer; Adenocarcinoma of the prostate; Sunitinib Malate; SUO11248; Sutent; BMS-354825; Sprycel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Sunitinib; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Abiraterone Acetate + Prednisone (AP) (Experimental): Abiraterone Acetate at 1000 mg orally each day, given in combination with 5 mg of Prednisone orally twice daily.
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone
- Group 1: AP + Sunitinib (Experimental): AP (Abiraterone Acetate + Prednisone) Plus Sunitinib; Randomized from AP group to receive Sunitinib if disease worsens. Assignment to crossover group AP + Dasatinib with further disease progression.
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone; Drug: Sunitinib
- Group 2: AP + Dasatinib (Experimental): AP (Abiraterone Acetate + Prednisone) Plus Dasatinib; Randomized from AP group to receive Dasatinib if disease worsens. Assignment to crossover group AP + Sunitinib with further disease progression.
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone; Drug: Dasatinib

INTERVENTIONS:
Drug: Abiraterone Acetate — 1000 mg by mouth each day of a 28 day cycle.
  Other Names: CB7630
Drug: Prednisone — 5 mg by mouth twice daily of a 28 day cycle.
Drug: Sunitinib — 37.5 mg by mouth daily for two weeks followed by a week of rest in a 28 day cycle.
  Other Names: Sunitinib Malate; SUO11248; Sutent
  Arms: Group 1: AP + Sunitinib
Drug: Dasatinib — 100 mg by mouth each day of a 28 day cycle.
  Other Names: BMS-354825; Sprycel
  Arms: Group 2: AP + Dasatinib

SUMMARY:
You are being asked to take part in this study because you have prostate cancer that has spread to other parts of the body.

This is an investigational study. Prednisone is FDA-approved and commercially available. Abiraterone acetate is FDA-approved and commercially available, but is still being researched. Sunitinib malate is FDA-approved for the treatment of gastrointestinal tumors and renal cell carcinoma, and dasatinib is FDA approved and commercially available for certain types of leukemia. The use of these drugs in prostate cancer and in combination with abiraterone acetate and prednisone is investigational.

Up to 180 patients will be enrolled in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
The Study Drugs:

Abiraterone acetate is designed to block male hormones in the body that may cause prostate cancer to grow.

Prednisone is commonly given in combination with other drugs to patients with prostate cancer. In this study, it is being used in combination with abiraterone acetate in order to help prevent side effects that abiraterone acetate may cause.

Sunitinib malate is designed to block pathways that control important events such as the growth of blood vessels that are essential for the growth of cancer.

Dasatinib is designed to change the function of genes. By changing the function of these genes, it may prevent cancer from growing and spreading.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take 4 tablets of abiraterone acetate by mouth every day. The tablets should be taken all at once, at least 1 hour before a meal or 2 hours after a meal. You will also take 1 tablet of prednisone by mouth 2 times each day. You will take both of these drugs throughout the entire study.

If the disease gets worse while you are taking abiraterone acetate and prednisone, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups.

* If you are assigned to Group 1, you will start taking sunitinib malate. You will take 3 capsules by mouth 1 time each day, while continuing to take abiraterone acetate and prednisone.
* If you are assigned to Group 2, you will start taking dasatinib. You will take 2 tablets by mouth 1 time each day, while continuing to take abiraterone acetate and prednisone. Dasatinib tablets should be swallowed whole, with or without a meal. If you accidentally miss taking a dose of dasatinib, it may be taken within 12 hours later. If you vomit within 30 minutes of taking the tablets, that dose may be repeated. If you miss a dose due to side effects, the dose should not be replaced.

If the disease gets worse after you have been assigned to a group, and you are still eligible to continue taking the study drugs, you will "crossover" to the other group. If you were in Group 1, you would stop taking sunitinib malate and begin taking dasatinib. If you were in Group 2, you would stop taking dasatinib and begin taking sunitinib malate. No matter which group you crossover to, you will continue taking abiraterone acetate and prednisone.

Study Visits:

At each study visit, you will be asked about any other drugs you may be receiving and about any side effects you may be having.

Every 2 weeks during the first 12 weeks of taking abiraterone acetate and prednisone and during the first 3 cycles (9-12 weeks) of each new treatment combination, blood (about 1-2 tablespoons) will be collected to test your liver function.

Every 4 weeks, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* Blood (about 1-2 tablespoons) and urine will be collected for routine tests. Part of this blood will be used to measure your PSA and your levels of a specific marker of prostate cancer.
* You will be asked questions about how you are feeling and about any side effects you may have had since your last visit.
* You will be asked about any other drugs you may be taking.
* Your performance status will be recorded.

If the disease gets worse (or you change treatments) at any point in the study, the following tests and procedures will be performed:

* Blood (about 1-2 tablespoons) and urine will be collected for routine tests.
* You will have a bone marrow aspiration and biopsy or a tumor tissue biopsy to collect tumor tissue from places to which the tumor has spread to check the status of the disease.
* You will have an ECG and an echocardiogram or a MUGA scan.
* You will have a chest x-ray, CT scans of your abdomen and pelvis, and a bone scan to check the status of your disease.

If your doctor thinks it is necessary:

°You will have a chest x-ray, CT scans of your abdomen and pelvis, and a bone scan to check the status of your disease.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will be taken off study if the disease gets worse after crossover, if you experience intolerable side effects, or if the doctor thinks that it is in your best interest.

End of Treatment Visit:

After you stop receiving the study drugs for any reason, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* Blood (about 1-2 tablespoons) will be drawn for routine tests and to check your PSA level, your level of a specific marker of prostate cancer, and to check for a protein related to cancer.
* You will be asked questions about how you are feeling and about any side effects you may have had since your last visit.
* You will be asked about any other drugs you may be taking.
* Your performance status will be recorded.
* You will have a bone marrow aspiration and biopsy or a tumor tissue biopsy to collect tumor tissue from places to which the tumor has spread to check the status of the disease.

Post-Treatment (Safety) Follow-Up Visit:

About 30 days after your last dose of study drugs, the following tests and procedures will be performed:

* You will have a physical exam, including a measurement of your vital signs.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* Your performance status will be recorded.
* You will be asked about any side effects you may have experienced since your last visit.
* You will be asked about any other drugs you may be taking.

Long-Term Follow-Up:

A member of the study staff will check up on you about every 6 months after your Post-Treatment (Safety) Follow-Up Visit. This will consist of a phone call, an e-mail, or a review of your medical and/or other records. If you are contacted by phone, the call will only last a few minutes.

After your End-of-Treatment visit, the study staff will contact you by phone, e-mail, or you will come in for a clinic visit. You will be asked about how you are feeling and any side effects you may have had. Each follow-up will take about 5 minutes. Follow-up will take place every 3 months for the first 2 years, every 6 months for the third year, and 1 time a year after that. The last follow-up will be about 5 years after the last patient is enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Male aged 18 years and above
3. Histologically or cytologically confirmed adenocarcinoma of the prostate
4. Metastatic disease documented by positive bone scan or metastatic lesions other than liver or visceral metastasis on CT or MRI.
5. Prostate cancer progression documented by PSA according to PCWG2 or radiographic progression according to modified RECIST criteria
6. Surgically or medically castrated, with testosterone levels of </= 50 ng/dL (</= 2.0 nM). If the patient is being treated with LHRH agonists (patients who have not undergone orchiectomy), this therapy must have been initiated at least 4 weeks prior to Cycle 1 Day 1 and must be continued throughout the study.
7. If the patient received previous anti-androgen therapy, then they have shown progression after withdrawal. Patients who received combined androgen blockade with an anti-androgen must have shown PSA progression after discontinuing the anti-androgen prior to enrollment (>/= 4 weeks since last flutamide, >/= 6 weeks since last bicalutamide or nilutamide). If progression is documented prior to this time interval, patients are eligible.
8. Previous treatment with docetaxel is allowed. Patients must have recovered from any acute toxicity related to the treatment to be eligible.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of </= 1.
10. Hemoglobin >/= 9.0 g/dL
11. Platelet count >/= 100,000/microL
12. Serum albumin >/= 3.5 g/dL
13. Serum creatinine </= 1.5 x ULN or a calculated creatinine clearance >/= 60 mL/min
14. Serum potassium >/= 3.5 mmol/L
15. Serum sodium, magnesium, potassium, phosphate, and calcium >/= LLN (lower limit of normal)
16. ANC value >/= 1,000/mm^3
17. Liver function: i. Serum bilirubin </= 1.5 x ULN (except for patients with documented Gilbert's disease) ii. AST or ALT </= 2.5 x ULN
18. Able to swallow the study drug whole as a tablet/capsule.
19. Patients who have partners of childbearing potential (.e.g. female that has not been surgically sterilized or who are not amenorrheic for >/= 12 months) must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator during the study and for 13 weeks after last study drug administration.
20. Concomitant Medications (i) Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy (at least 5 days prior). (ii) Patient agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia; (iii) Patient agrees to discontinue use of drugs primarily metabolized by CYP3A4 enzyme; (iv) Patient agrees to discontinue use of H2 Inhibitors or proton inhibitors prior to dasatinib administration.

Exclusion Criteria:

1. Active infection (requiring oral or IV antibiotics) or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
2. Any chronic medical condition requiring a higher dose of corticosteroid than 5mg prednisone/prednisolone twice daily.
3. Pathological finding consistent with small cell carcinoma of the prostate
4. Radiation therapy for treatment of the primary tumor within 6 weeks of Cycle 1, Day 1. Patients who have received palliative radiation to a single site and recovered are eligible.
5. No malignancy [other than the one treated in this study] which required radiotherapy or systemic treatment within the past 5 years.)
6. Previously treated with ketoconazole (for prostate cancer) for greater than 7 consecutive days OR previously treated with any other -azole drug (e.g. fluconazole, itraconazole) within 4 weeks of Cycle 1, Day 1
7. Prior flutamide (Eulexin) treatment within 4 weeks of Cycle 1, Day 1 (patients whose PSA did not decline for three or more months in response to antiandrogen given as a second line or later intervention will require only a two week washout prior to Cycle 1, Day 1)
8. Bicalutamide (Casodex), nilutamide (Nilandron) within 6 weeks of Cycle 1 Day 1 (patients whose PSA did not decline for three or more months in response to antiandrogen given as a second line or later intervention will require only a two week washout prior to Cycle 1, Day 1)
9. Uncontrolled hypertension (systolic BP >/= 140 mmHg or diastolic BP >/= 90 mmHg). Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
10. Prolonged QTc interval on pre-entry electrocardiogram (>/= 450 msec)
11. Active or symptomatic viral hepatitis or chronic liver disease
12. History of pituitary or adrenal dysfunction
13. Known brain metastasis
14. Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes), Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 50% at baseline
15. History of significant bleeding disorder unrelated to cancer, including: i) Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease) ii) Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies) iii) Ongoing or recent (</= 3 months) significant gastrointestinal bleeding
16. Atrial fibrillation or other cardiac arrhythmia requiring digitalis
17. Other malignancy, except non-melanoma skin cancer, with a >/= 30% probability of recurrence within 24 months
18. Clinically significant pleural effusion as determined by the Principal Investigator.
19. Administration of an investigational therapy for prostate cancer within 30 days of Cycle 1, Day 1
20. Any condition which, in the opinion of the investigator, would preclude participation in this trial.
21. Patients taking category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib) i) quinidine, procainamide, disopyramide ii) amiodarone, sotalol, ibutilide, dofetilide iii) erythromycin, clarithromycin iv) chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide v) cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
22. Prisoners or subjects who are involuntarily incarcerated.
23. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2011-03-16 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Corn, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Sakellakis MJ, Hahn AW, Ramachandran S, Zhang M, Hoang A, Song JH, Liu J, Wang F, Basu HS, Sheperd P, Wang X, Frigo DE, Lin SH, Panaretakis T, Zhang J, Navone N, Troncoso P, Logothetis CJ, Titus MA. Characterization of prostate cancer adrenal metastases: dependence upon androgen receptor signaling and steroid hormones. Prostate Cancer Prostatic Dis. 2023 Dec;26(4):751-758. doi: 10.1038/s41391-022-00590-x. Epub 2022 Sep 13. PMID 36100698
- [Derived] Boukovala M, Spetsieris N, Weldon JA, Tsikkinis A, Hoang A, Aparicio A, Tu SM, Araujo JC, Zurita AJ, Corn PG, Pagliaro L, Kim J, Wang J, Subudhi SK, Tannir NM, Logothetis CJ, Troncoso P, Wen S, Efstathiou E. A candidate androgen signalling signature predictive of response to abiraterone acetate in men with metastatic castration-resistant prostate cancer. Eur J Cancer. 2020 Mar;127:67-75. doi: 10.1016/j.ejca.2019.12.027. Epub 2020 Jan 24. PMID 31986451
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2011 to February 2015, patients were recruited from the outpatient clinics of Genitourinay Medical Oncology at MD Anderson Cancer Center in Houston, TX who have been diagnosed with metastatic prostate cancer.
Pre-assignment Details: 190 subjects were assessed for eligibility however of those 190 subjects, 10 did not meet eligibility criteria and 1 declined participation. A total of 179 subjects started on trial and received Abiraterone Acetate + Prednisone (AP). Of the 179 subjects that started on trial, 132 were randomized to the combination arms (64 to AP + Sunitinib and 68 to AP + Dasatinib).
Groups:
- Abiraterone Acetate + Prednisone (AP): Abiraterone Acetate at 1000mg orally each day, given in combination with 5mg of Prednisone orally twice daily
- AP + Sunitinib: AP (Abiraterone Acetate + Prednisone) Plus Sunitinib; Randomized from AP group to receive Sunitinib if disease worsens. Assignment to crossover group AP + Dasatinib with further disease progression.
- AP + Dasatinib: AP (Abiraterone Acetate + Prednisone) Plus Dasatinib; Randomized from AP group to receive Dasatinib if disease worsens. Assignment to crossover group AP + Sunitinib with further disease progression.
Period: Abiraterone Acetate+Prednisone(AP) Phase
Arm/Group | Abiraterone Acetate + Prednisone (AP) | AP + Sunitinib | AP + Dasatinib
Started | 179 | 0 | 0
Randomized to AP + Sunitinib | 64 | 0 | 0
Randomized to AP + Dasatinib | 68 | 0 | 0
Crossover to AP + Sunitinib | 0 | 0 | 0
Crossover to AP + Dasatanib | 0 | 0 | 0
Completed | 132 | 0 | 0
Not Completed | 47 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 24 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Not completed — Non-compliance | 2 | 0 | 0
Not completed — Ongoing Response to Abiraterone | 7 | 0 | 0
Period: Randomization Phase
Arm/Group | Abiraterone Acetate + Prednisone (AP) | AP + Sunitinib | AP + Dasatinib
Started | 0 | 64 | 68
Crossover to AP + Sunitinib | 0 | 0 | 32
Crossover to AP + Dasatanib | 0 | 39 | 0
Completed | 0 | 31 | 22
Not Completed | 0 | 33 | 46
Not completed — Adverse Event | 0 | 5 | 17
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 20 | 25
Not completed — Withdrawal by Subject | 0 | 4 | 2
Not completed — Non-Compliance | 0 | 1 | 0
Not completed — Comorbidities | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Of the 179 subjects that started on trial, 132 were randomized to the combination arms (64 to AP + Sunitinib and 68 to AP + Dasatinib).
Groups:
- Total: Total of all reporting groups
Arm/Group | Abiraterone Acetate + Prednisone (AP) | AP + Sunitinib | AP + Dasatinib | Total
Number analyzed (Participants) | 179 | 0 | 0 | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 84 |  |  | 84
  >=65 years | 95 |  |  | 95
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  |  | 0
  Male | 179 |  |  | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 |  |  | 25
  Not Hispanic or Latino | 58 |  |  | 58
  Unknown or Not Reported | 96 |  |  | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 3 |  |  | 3
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 19 |  |  | 19
  White | 146 |  |  | 146
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 11 |  |  | 11
Region of Enrollment [Number; unit: participants]
  United States | 179 |  |  | 179

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure (TTF)
Description: Time to treatment failure (TTF), defined as time from randomization (AP+S or AP+D) to progression per PCWG2 criteria or death.
Time Frame: Up to 11 months
Population: The first group/arm was not reported as the outcome measure of time to treatment failure is defined as the time from randomization (subjects were randomized after being in the first group/arm) to progression.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate + Prednisone (AP) | AP + Sunitinib | AP + Dasatinib
Number analyzed (Participants) | 0 | 64 | 68
Months |  | 5.5 [4.6 to 6.8] | 5.7 [3.8 to 7.4]

ADVERSE EVENTS:
Time Frame: Monitored continuously from baseline/first dose until 30 days post last dose, an average of 1 year
Description: •Death • A Life-threatening adverse drug experience-it does not include an adverse experience that might have caused death •Inpatient hospitalization or prolongation of existing hospitalization •A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions •A congenital anomaly/birth defect. The AEs are identified based on the arms the subjects were in. Each column is titled to show what study drug the subject was on when the AE occurred.
Groups:
- AP + Sunitinib → AP + Dasatanib: Randomized from AP group to receive AP + Sunitinib now on crossover group to receive AP + Dasatinib due to further disease progression.
- AP + Dasatanib → AP + Sunitinib: Randomized from AP group to receive AP + Dasatanib now on crossover group to receive AP + Sunitinib due to further disease progression.
Arm/Group | Abiraterone Acetate + Prednisone (AP) | AP + Sunitinib | AP + Sunitinib → AP + Dasatanib | AP + Dasatinib | AP + Dasatanib → AP + Sunitinib
All-Cause Mortality (participants affected / at risk) | 0/179 | 1/64 | 0/39 | 0/68 | 0/32
Serious Adverse Events (participants affected / at risk) | 8/179 | 11/64 | 0/39 | 10/68 | 0/32
Other Adverse Events (participants affected / at risk) | 46/179 | 33/64 | 31/39 | 43/68 | 24/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate + Prednisone (AP) (N=179) | AP + Sunitinib (N=64) | AP + Sunitinib → AP + Dasatanib (N=39) | AP + Dasatinib (N=68) | AP + Dasatanib → AP + Sunitinib (N=32)
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | NA | 0 | NA
Diarrhea (Gastrointestinal disorders) | 1 | 0 | NA | 0 | NA
Dehydration (Metabolism and nutrition disorders) | 2 | 4 | NA | 0 | NA
Facial Pain (General disorders) | 1 | 0 | NA | 0 | NA
Fever (General disorders) | 2 | 0 | NA | 1 | NA
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | 0 | NA
Lung Infection (Infections and infestations) | 1 | 0 | NA | 0 | NA
Chest Pain-Cardiac (Cardiac disorders) | 1 | 0 | NA | 0 | NA
Cardiac disorders- other (Cardiac disorders) | 0 | 1 | NA | 2 | NA
Hematuria (Renal and urinary disorders) | 0 | 2 | NA | 0 | NA
Spinal Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | 0 | NA
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | NA | 1 | NA
Syncope (Nervous system disorders) | 0 | 2 | NA | 0 | NA
Fall (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | 0 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | NA | 1 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | NA | 1 | NA
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | NA | 1 | NA
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | NA | 1 | NA
Dizziness (Nervous system disorders) | 0 | 0 | NA | 1 | NA
Headaches (Nervous system disorders) | 0 | 0 | NA | 1 | NA
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | NA | 2 | NA
Surgical and medical procedures - other (Surgical and medical procedures) | 0 | 0 | NA | 1 | NA
Urinary Tract Infection (Infections and infestations) | 0 | 0 | NA | 1 | NA
Sepsis (Infections and infestations) | 0 | 0 | NA | 1 | NA
Myocardial Infarction (Cardiac disorders) | 0 | 0 | NA | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate + Prednisone (AP) (N=179) | AP + Sunitinib (N=64) | AP + Sunitinib → AP + Dasatanib (N=39) | AP + Dasatinib (N=68) | AP + Dasatanib → AP + Sunitinib (N=32)
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 0 | 4 | 2
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 0 | 2 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 11 | 9 | 10 | 12 | 7
Alkaline Phosphatase Increased (Investigations) | 23 | 16 | 22 | 24 | 15
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0
Anemia (Blood and lymphatic system disorders) | 42 | 27 | 28 | 37 | 19
Anorexia (Metabolism and nutrition disorders) | 0 | 3 | 7 | 9 | 7
Anxiety (General disorders) | 6 | 0 | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 0 | 3
Aspartate Aminotransferase Increased (Investigations) | 16 | 12 | 16 | 15 | 13
Back Pain (Musculoskeletal and connective tissue disorders) | 20 | 25 | 17 | 23 | 15
Blood Bilirubin Increased (Investigations) | 7 | 10 | 3 | 7 | 7
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6 | 5
Bruising (General disorders) | 0 | 4 | 2 | 4 | 3
Cardiac disorders - other (Cardiac disorders) | 0 | 0 | 3 | 0 | 0
Cholesterol high (Investigations) | 0 | 0 | 2 | 0 | 3
Constipation (Gastrointestinal disorders) | 11 | 6 | 12 | 11 | 12
COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 9 | 9 | 5
Creatinine Increased (Investigations) | 9 | 8 | 7 | 13 | 4
Depression (General disorders) | 8 | 4 | 3 | 8 | 0
Diarrhea (Gastrointestinal disorders) | 8 | 16 | 18 | 12 | 12
Dizziness (Nervous system disorders) | 0 | 8 | 2 | 4 | 5
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 0 | 4
Dysesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 10 | 12 | 6 | 11
Dyspepsia (Gastrointestinal disorders) | 0 | 7 | 7 | 5 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 14 | 18 | 7
Edema Face (General disorders) | 0 | 0 | 3 | 0 | 0
Edema Limbs (General disorders) | 13 | 7 | 15 | 19 | 5
Eye disorders - other (Eye disorders) | 0 | 3 | 0 | 0 | 0
Fatigue (General disorders) | 29 | 26 | 29 | 38 | 21
Fever (General disorders) | 0 | 3 | 3 | 5 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 4 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 3 | 4 | 0 | 4
Gastrointestinal disorders - other (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 0 | 2
Headache (Nervous system disorders) | 0 | 5 | 7 | 8 | 7
Hematuria (Renal and urinary disorders) | 0 | 3 | 7 | 4 | 5
Hemoglobinuria (Renal and urinary disorders) | 0 | 4 | 7 | 0 | 0
Hot Flashes (Vascular disorders) | 19 | 19 | 12 | 20 | 14
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 4 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 15 | 10 | 12 | 10 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 3 | 3 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 7 | 0 | 5 | 2
Hypertension (Vascular disorders) | 18 | 11 | 17 | 18 | 15
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 5 | 3 | 6 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 7 | 5 | 9 | 3
Hypokalemia (Metabolism and nutrition disorders) | 15 | 11 | 18 | 18 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 10 | 9 | 13 | 9 | 8
Hyponatremia (Metabolism and nutrition disorders) | 9 | 4 | 6 | 6 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 4 | 3 | 5 | 2
Hypotension (Vascular disorders) | 0 | 4 | 0 | 0 | 0
Infections and infestations - other (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Insomnia (General disorders) | 11 | 5 | 6 | 6 | 0
Lymphocyte count decreased (Investigations) | 0 | 4 | 3 | 5 | 6
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Mucositis Oral (Gastrointestinal disorders) | 0 | 6 | 9 | 0 | 6
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 0 | 2
Nausea (Gastrointestinal disorders) | 16 | 16 | 20 | 14 | 11
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 9 | 10 | 0 | 3
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 3 | 0 | 0
Oral Dysesthesia (General disorders) | 0 | 0 | 2 | 0 | 0
Oral Pain (General disorders) | 0 | 0 | 3 | 0 | 0
Pain (General disorders) | 32 | 24 | 26 | 29 | 17
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3 | 4 | 2
Palmar-Plantar Erythrodysesthesia Syndrom (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 0 | 2
Paresthesia (Nervous system disorders) | 0 | 3 | 4 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 3 | 4 | 6 | 3
Platelet Count Decreased (Investigations) | 0 | 10 | 7 | 6 | 6
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4
Proteinuria (Renal and urinary disorders) | 0 | 0 | 5 | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 4 | 5
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0
Skin Hipopigmentation (Skin and subcutaneous tissue disorders) | 0 | 5 | 8 | 0 | 2
Stomach Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Thromboembolic Event (Vascular disorders) | 0 | 0 | 3 | 0 | 0
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 0
Urinary Frequency (Renal and urinary disorders) | 19 | 11 | 11 | 16 | 9
Urinary Incontinence (Renal and urinary disorders) | 0 | 8 | 2 | 5 | 2
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 7 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 10 | 6 | 2
Weight Gain (Investigations) | 0 | 5 | 0 | 0 | 0
Weight Loss (Investigations) | 0 | 0 | 0 | 0 | 2
White Blood Cell Decreased (Investigations) | 0 | 15 | 11 | 5 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT01254864/Prot_SAP_000.pdf